CLINICAL TRIAL: NCT05038371
Title: Connective Tissue Growth Factor in Patients With Neovascular Age Related Macular Degeneration
Status: Terminated | Type: Observational
Why Stopped: The study team decided to not publish a manuscript therefore we decided to terminate the study
Sponsor: Johns Hopkins University (Other)
Collaborators: Olix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00255963
Record Dates: First submitted 2021-09-03; First posted 2021-09-09 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will only be used for measurement of biomarkers mentioned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with neovascular age-related macular degeneration: This will include 10 subjects with a diagnosis of age-related macular degeneration.
- Controls: This group will comprise 10 participants who plan to undergo vitrectomy for macular hole, macular pucker, or vitreomacular traction, vitreous floaters or another condition unrelated to scarring.

SUMMARY:
Age-related macular degeneration (AMD) remains a leading cause of blindness in United States and can be broadly divided into two forms: non-neovascular AMD (NNVAMD) and neovascular AMD (NVAMD) AMD. Among the several mechanisms underlying AMD, hypoxia and oxidative stress have been implicated and cause upregulation of several signaling proteins. About 20% of patients with NNVAMD develop choroidal neovascularization and hence convert to NVAMD. Upregulation of vascular endothelial growth factor (VEGF) plays a critical role in conversion from NNVAMD to NVAMD.

Connective tissue growth factor (CTGF) is a polypeptide that has been shown to be overexpressed in various fibrotic disorders, suggesting its involvement in scarring. After the development of choroidal neovascularization, subretinal fibrosis may occur and result in permanent reduction of vision. An important question is, does CTGF contribute to subretinal fibrosis. An important first step in addressing this question is to determine if CTGF levels are increased in the eyes of patients with NVAMD and this is the objective of this study.

The investigators plan to measure levels of connective tissue growth factor (CTGF) in the aqueous humor of patients with neovascular age-related macular degeneration and compare to controls. Levels of VEGF will be measured as a positive control.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Willing to sign informed consent and authorization of use and disclosure of protected health information
* For study group: patients must have a clinical diagnosis of NVAMD
* For control group: patients undergoing vitrectomy for macular hole, macular pucker, or vitreomacular traction, vitreous floaters or another condition unrelated to scarring.

Exclusion Criteria:

* Subjects with a retinal condition other than NVAMD in which scarring may occur such as proliferative vitreoretinopathy or retinal detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of twenty eligible patients, 10 with NVAMD and 10 controls will be enrolled.
  Patients and controls will be identified and recruited through the clinic population of co-investigators at the Wilmer Eye Institute.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Measurement of aqueous humor levels of CTGF by ELISA | Baseline visit
  Connective tissue growth factor (CTGF) levels will be measured, using ELISA, in aqueous samples of both patients and controls.
Measurement of aqueous humor levels of VEGF by ELISA | Baseline visit
  Vascular endothelial growth factor (VEGF) levels will be measured, using ELISA, in aqueous samples of both patients and controls. Levels of VEGF will serve as a positive control.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, M.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No